CLINICAL TRIAL: NCT00411736
Title: Supplementary Oral Azithromycin in Treatment of Intermittent Pseudomonas Aeruginosa Colonization in CF-patients With Inhaled Colistin and Oral Ciprofloxacin; Postponing Next Isolate of Pseudomonas and Prevention of Chronic Infection. A Prospective, Double-blinded, Placebo-controlled Scandinavian Multi-centre Study.
Brief Title: Scandinavian Cystic Fibrosis Azithromycin Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Christine Hansen, Medical doctor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AZI/SCAND/01
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Pseudomonas aeruginosa; Azithromycin; Intermittent pulmonary infection
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Stratification group: Age under 8 years, no CF siblings at home.
  Interventions: Drug: Study medication, azithromycin or placebo
- B (Experimental): Stratification group: Age >/= 8 years, no CF siblings at home.
  Interventions: Drug: Azithromycin or placebo tablets
- C (Experimental): Stratification group: Age >/= 8 years, CF siblings at home.
  Interventions: Drug: Azithromycin or placebo tablets

INTERVENTIONS:
Drug: Study medication, azithromycin or placebo — Granulate for syrup in the group under 8 years, 40 mg/ml. Dose: 5 mg/kg/day in one daily dose.
  Other Names: Projectnumber HSA06-20/1
  Arms: A
Drug: Azithromycin or placebo tablets — Tablets of 250 mg, azithromycin or placebo. Dosage: 1 tablet every other day for participants with a weight less than 40 kg´s. 1 tablet every day for participants weighing 40 kg´s or more.
  Other Names: Project number HSA06-20/1
  Arms: B; C

SUMMARY:
In patients with Cystic Fibrosis, recurrent airway infection caused by Pseudomonas aeruginosa ultimately leads to chronic airway infection. The purpose of this study is to determine whether supplementary low-dose azithromycin to standard inhaled colistin and oral ciprofloxacin in the treatment of intermittent pseudomonas airway-infection can postpone the next episode of intermittent pseudomonas airway-infection and prevent development of chronic airway-infection.

DETAILED DESCRIPTION:
Cystic Fibrosis is the most common genetic, inherited, deadly disease in caucasians. The disease is characterized by recurrent airway-infections caused by Pseudomonas aeruginosa, ultimately leading to chronic airway-infection, which is the main cause of the increased morbidity and mortality seen in this disease.

P. aeruginosa has the ability to change to mucoid phenotype - producing alginate and growing in biofilm, which protects the microorganisms from antibiotics and leukocytes. The change in phenotype is seen as chronic infection is established and eradication becomes impossible. Treatment with long-term, low-dose azithromycin in chronically infected CF-patients can improve the clinical condition of the patients. The exact mechanism for this is not known, but is possibly a combination of anti-inflammatory effects and the ability of azithromycin to inhibit alginate-production. Inhibition of biofilm-formation leaves the bacteria more susceptible to the actions of antibiotics and leukocytes.

Prior to establishment of chronic infection, recurrent, intermittent colonization of the airways with non-mucoid P. aeruginosa is seen. Intermittent infections can be treated using a combination of antibiotics, thereby postponing the next episode of airway-infection with P. aeruginosa.

The purpose of this study is to clarify wether supplementary azithromycin in the treatment of intermittent pseudomonas-infection in CF-patients can lead to further postponement of next pseudomonas-colonization and maybe prevent development of chronic infection. This is done in a randomised, double-blinded, placebo-controlled multicentre study.

2 treatments will be compared:

1. Inhaled colistin and oral ciprofloxacin in combination with oral azithromycin
2. Inhaled colistin and oral ciprofloxacin in combination with oral placebo.

The treatment will be given for 3 weeks, and the primary end-point is the time until next colonization with P. aeruginosa in the airways of the patients, comparing the 2 treatment-groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis based on genotype and/or positive sweat-test
* Written informed consent based on written and spoken information
* No chronic airway-infections with Gram-negative bacteria
* Fertile, sexually active women must use contraception (p-pills, IUD or other methods with a similar Pearl-index) when participating in the study

Exclusion Criteria:

* P. aeruginosa in airway secretions obtained less than 3 months prior to inclusion
* Chronic infection of the airways caused by Gram-negative bacteria (Burkholderia species, Achromobacter xylosoxidans, Pandorea apista or Stenotrophomonas maltophilia)
* Chronic infection of the airways caused by P. aeruginosa (chronic infection is defined by continuing growth of the microorganism for 6 months and/or an increase in specific, precipitating antibodies to a level of at least 2)
* Previous infection with a strain of P. aeruginosa resistant to ciprofloxacin or colistin
* Previous participation in a pseudomonas-vaccination-study
* Patients younger than 1 year
* Pregnant or lactating women, or sexually active women unwilling to use safe contraception (p-pills, IUD or method with similar Pearl-index) when participating in the study
* Severe insufficiency of the liver or kidneys as judged by the local investigator

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-05; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Time to next airway-colonization (re-colonization) with Pseudomonas aeruginosa | up to 5 years

SECONDARY OUTCOMES:
Clinical condition of the patients (height, weight and lung function) | up to 5 years
Bacteriological examination of Pseudomonas aeruginosa (phenotype, resistance) | 5 years
Genotyping of Pseudomonas aeruginosa using Pulsed Field Gel Electrophoresis (re-infection caused by identical or new strain) | 5 years
Specific, precipitating pseudomonas-antibodies (establishment of chronic infection) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Niels Hoiby, Prof.M.D.DSc, Principal Investigator — Department of Clinical Microbiology, Rigshospitalet
Locations (8):
- Denmark (2):
  - CF-centre Skejby, Skejby Sygehus, Brendstrupgaardsvej 100, Aarhus N
  - CF-centre Copenhagen, Rigshospitalet, Blegdamsvej 9, Copenhagen
- Norway (2):
  - CF-centre Bergen, Haukeland Universitetssykehus, Bergen
  - CF-centre Oslo, Ullevaal Universitetssykehus, Oslo
- Sweden (4):
  - CF-centre Göteborg, Drottning Silvias barn- och ungdomssjukhus, Gothenburg
  - CF-centre Lund, Universitetssjukhuset i Lund, Lund
  - CF-centre Stockholm, Karolinska Universitetssjukhuset, Huddinge, Stockholm
  - CF-centre Uppsala, Akademiska Barnsjukhuset, Uppsala

REFERENCES:
- [Background] Doring G, Conway SP, Heijerman HG, Hodson ME, Hoiby N, Smyth A, Touw DJ. Antibiotic therapy against Pseudomonas aeruginosa in cystic fibrosis: a European consensus. Eur Respir J. 2000 Oct;16(4):749-67. doi: 10.1034/j.1399-3003.2000.16d30.x. PMID 11106223
- [Background] Hoiby N, Frederiksen B, Pressler T. Eradication of early Pseudomonas aeruginosa infection. J Cyst Fibros. 2005 Aug;4 Suppl 2:49-54. doi: 10.1016/j.jcf.2005.05.018. PMID 16023416
- [Background] Valerius NH, Koch C, Hoiby N. Prevention of chronic Pseudomonas aeruginosa colonisation in cystic fibrosis by early treatment. Lancet. 1991 Sep 21;338(8769):725-6. doi: 10.1016/0140-6736(91)91446-2. PMID 1679870
- [Background] Equi A, Balfour-Lynn IM, Bush A, Rosenthal M. Long term azithromycin in children with cystic fibrosis: a randomised, placebo-controlled crossover trial. Lancet. 2002 Sep 28;360(9338):978-84. doi: 10.1016/s0140-6736(02)11081-6. PMID 12383667
- [Background] Gillis RJ, White KG, Choi KH, Wagner VE, Schweizer HP, Iglewski BH. Molecular basis of azithromycin-resistant Pseudomonas aeruginosa biofilms. Antimicrob Agents Chemother. 2005 Sep;49(9):3858-67. doi: 10.1128/AAC.49.9.3858-3867.2005. PMID 16127063
- [Background] Hansen CR, Pressler T, Koch C, Hoiby N. Long-term azitromycin treatment of cystic fibrosis patients with chronic Pseudomonas aeruginosa infection; an observational cohort study. J Cyst Fibros. 2005 Mar;4(1):35-40. doi: 10.1016/j.jcf.2004.09.001. PMID 15752679
- [Background] Jaffe A, Francis J, Rosenthal M, Bush A. Long-term azithromycin may improve lung function in children with cystic fibrosis. Lancet. 1998 Feb 7;351(9100):420. doi: 10.1016/S0140-6736(05)78360-4. No abstract available. PMID 9482305
- [Background] Saiman L, Marshall BC, Mayer-Hamblett N, Burns JL, Quittner AL, Cibene DA, Coquillette S, Fieberg AY, Accurso FJ, Campbell PW 3rd; Macrolide Study Group. Azithromycin in patients with cystic fibrosis chronically infected with Pseudomonas aeruginosa: a randomized controlled trial. JAMA. 2003 Oct 1;290(13):1749-56. doi: 10.1001/jama.290.13.1749. PMID 14519709
- [Background] Wolter J, Seeney S, Bell S, Bowler S, Masel P, McCormack J. Effect of long term treatment with azithromycin on disease parameters in cystic fibrosis: a randomised trial. Thorax. 2002 Mar;57(3):212-6. doi: 10.1136/thorax.57.3.212. PMID 11867823
- [Background] Kobayashi H. Biofilm disease: its clinical manifestation and therapeutic possibilities of macrolides. Am J Med. 1995 Dec 29;99(6A):26S-30S. doi: 10.1016/s0002-9343(99)80282-4. PMID 8585531